CLINICAL TRIAL: NCT07259460
Title: Effects of Dexmedetomidine Delivered With Target Controlled Infusion (TCI) on Patient State Index Values, Electroencephalographic Spectrum, Analgesia Nociception Index nd Pupillomtry Values During Total Intravenous Anesthesia With Propofol TCI
Brief Title: Effects of Dexmedetomidine Target Controlled Infusion on Patient State Index Values and Electroencephalographic Spectrum During Total Intravenous Anesthesia With Propofol
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, PhD, Principal investigator, University of Padova
Other Study IDs: DexMAST
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Adjuvants, Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dexmedetomidine Target Controlled infusion (TCI, Dyck model) effects on Neuromonitoring during Total Intravenous Anesthesia (TIVA) with Propofol and Remifentanil TCI (Eleveld model) has not been investigate yet.

Authors aim to investigate its effect on Patient State index (PSi), the power spectrum EEG, the Analgesia Nociception Index (ANI) and pupillometry values during maintenance during TIVA-TCI with Propofol, Remifentanil and Dexmedetomidine.

DETAILED DESCRIPTION:
The effects of Dexmedetomidine administered via Target-Controlled Infusion (TCI, Dyck model) on neuromonitoring during Total Intravenous Anesthesia (TIVA) with Propofol and Remifentanil (TCI, Eleveld model) have not yet been investigated.

The authors aim to systematically evaluate the impact of adding Dexmedetomidine on key neuromonitoring parameters commonly used in clinical anesthesia during the maintenance phase of TIVA-TCI. Specifically, the study will assess:

Patient State Index (PSi) as a measure of the hypnotic state;

Electroencephalographic (EEG) power spectrum, to identify changes in cortical activity patterns associated with Dexmedetomidine administration;

Analgesia Nociception Index (ANI), to evaluate potential modifications in the analgesia-nociception balance;

Pupillometry, to quantify autonomic and pupillary responses to stimuli.

This investigation aims to determine whether the addition of Dexmedetomidine using a TCI approach produces predictable and clinically relevant alterations in neurophysiological monitoring during anesthesia with Propofol and Remifentanil. Ultimately, the study seeks to support more precise drug titration and enhance patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol and Rmifntanil (Eleveld model) and Dexmedetomidine (Dyck model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity
* Regional anesthesia performed

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol, remifentanil and Dexmedetomidine TCI will be recruited
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Dexmedetomidine on Patient State index (PSi) during stable Propofol - Remifentanil general anesthesia | PSi values and DexmedetomidineTarget Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if Dexmedetomidine variations during general anesthesia has an impact on the PSi values
Effects of Dexmedetomidine on Electroencephalogram (EEG) power spectrum during stable Propofol - remifentanil general anesthesia | EEG power spectrum and DexmedetomidineTarget Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if dexmedetomidine variations during general anesthesia has an impact on the EEG power spectrum
Effects of Dexmedetomidine on Analgesia Nociception Index (ANI) during stable Propofol general anesthesia | ANI values and Sufentanil Target Controlled Infusion (TCI) concentrations will be monitored during all the time of surgery
  Evaluate if dxmedetomidine variations during general anesthesia has an impact on the ANI values

SECONDARY OUTCOMES:
Analgesia Nociception Index (ANI) values and postoperative pain | Numeric Rating Scale (NRS) will be evaluated after the end of surgery and 24 hours after the end of surgery and compared to ANI values after 24 hours
  Evaluate if different ANI values at the same dexmedetomidine concentrations has an impact on postoperative pain
Patient State Index (PSi) values and postoperative delirium | Confusion assessment method (CAM) test for delirium will be performed after the end of surgery and compared to PSi values after 24 hours
  Evaluate if different PSi values at the same dexmedetomidine concentrations has an impact on postoperative delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy

IPD SHARING:
Plan to Share IPD: Undecided